CLINICAL TRIAL: NCT03886441
Title: A Randomized, Open Phase II Study of the Incidence and Safety of Radiation Pneumonia in Patients With Locally Advanced NSCLC Treated With Beclomethasone Propionate Inhaled During Radical Radiotherapy Compared With Conventional Radiotherapy
Brief Title: Prevention of Locally Advanced NSCLC Radiotherapy Pneumonia by Inhaling Beclomethasone Propionate
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tongji University (Other)
Collaborators: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Caicun Zhou, Professor, doctor, Tongji University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: fk1416
Record Dates: First submitted 2019-03-14; First posted 2019-03-22 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Locally Advanced Non Small Cell Lung Cancer
Keywords: beclomethasone propionate; radiation pneumonitis; NSCLC; radical radiotherapy; Preventive effect
MeSH Terms: conditions — Radiation Pneumonitis | interventions — beclomethasone 17-monopropionate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prevention group (Experimental): Participants inhaled beclomethasone propionate aerosol daily during chest radical radiotherapy (total dose 60GY).
  Interventions: Drug: Beclomethasone propionate
- Traditional therapy group (No Intervention): Participants were not given daily inhalation of beclomethasone propionate when undergoing radical chest radiotherapy (total dose 60GY).

INTERVENTIONS:
Drug: Beclomethasone propionate — Beclomethasone propionate inhaled twice daily during radiotherapy
  Arms: Prevention group

SUMMARY:
Radical radiotherapy is the main treatment of locally advanced lung cancer, and radiation pneumonia is the main toxic effects of radiotherapy. Among them, the fatality rate of severe radiation pneumonia can reach 50%, which is very harmful to tumor patients. At present, the treatment mode of radiation pneumonia is very few, and the therapeutic effect is poor. The prevention of radiation pneumonitis may be the best way to reduce the number of patients with Post-radiotherapy pneumonia. Previous small clinical studies have shown that the incidence of radiation pneumonia in inhaled beclomethasone group (2 /28) was significantly lower than that in oral prednisone group (8 /29) during radiotherapy. The purpose of this study was to compare the efficacy and safety of radiotherapy between the therapeutic group (inhaled beclomethasone during radiotherapy) and the control radiotherapy group (patients received radiotherapy only), especially the incidence of radiation-induced pneumonia within half a year.

DETAILED DESCRIPTION:
To compare the incidence of radiation pneumonia, effect and side effects of radiotherapy in lung between beclomethasone inhalation therapeutic group and control radiotherapy group in patients with locally advanced non-small cell lung cancer (NSCLC) during radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects understood the requirements and risks of the study fully and signed the informed consent form.
2. Aged between 18 and 70 years;
3. Histologically or cytologically confirmed diagnosis of locally advanced non-small cell lung cancer.
4. All of these patients have pointers to radical radiation and can't be treated surgically.
5. ECOG PS of 0-2;
6. Women of childbearing age had negative pregnancy tests and were willing to accept drugs or intrauterine contraception, while men of childbearing age were willing to accept contraception voluntarily.
7. Adequate hematologic function:

   Peripheral blood neutrophil count > 2000 cells / uL, Platelet count > 100*109 / L; Hemoglobin >9.0g/dL;
8. Blood total bilirubin < 2 times normal upper limit, blood AST and ALT ≤ 2. 5 times normal upper line;
9. Inosine clearance ≥ 60ml / min;
10. Life expectancy of at least 12weeks.

Exclusion Criteria:

1. With severe or uncontrolled systemic diseases;
2. With a history of asthma, systemic immune diseases, such as the need for long-term hormone treatment in patients;
3. The lung function decreased obviously;
4. Those receiving targeted therapy or biological therapy at the same time;
5. Allergic to beclomethasone propionate;
6. Pregnant or lactating women;
7. Accompanied by uncontrolled diabetes, need to take oral hormone treatment of sarcoidosis and vasculitis, lupus erythematosus and other immune diseases;
8. In recent 5 years has suffered from other tumors: cervical cancer, basal cell carcinoma of the skin, and so on;
9. The estimated survival time was less than 3 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of radiation pneumonia between two groups of patients | Chest CT assessment every 6 weeks since thoracic irradiation, up to 36 weeks.
  To evaluate the incidence of radiation pneumonia in 36weeks since thoracic irradiation between two groups of patients

SECONDARY OUTCOMES:
Objective Response Rate between two groups of patients | tumor assessment every 6 weeks since thoracic irradiation , up to 36 weeks.
  To evaluate Objective response rate every 6weeks since thoracic irradiation.
Side effects between two groups of patients | 36 weeks .
  To evaluated in the 36 weeks since the thoracic irradiation began according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0

OTHER OUTCOMES:
Quality of life between two groups of patients | 36 weeks
  evaluated every 6 weeks since the thoracic irradiation began according to the EORTC Quality-of-Life Questionnarire-Lung Cancer 13 Module(EORTC OLO-LC13)

CONTACTS AND LOCATIONS:
Overall Officials: caicun zhou, phD MD, Principal Investigator — Shanghai Pulmonary Hospital, Tongji University
Locations (1):
- Medical Department, Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China